CLINICAL TRIAL: NCT07103213
Title: Effectiveness of a School-based Programme Integrating Social Media Literacy and Third-wave Cognitive-behavioral Interventions in Promoting Positive Body Image Among Adolescents: a Cluster Randomized Controlled Trial
Brief Title: A School Program for Teenagers to Promote Positive Body Image Using Social Media Education and Self-Compassion-Based Activities
Acronym: IMPACTREEL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Sheila Fernández García, Maria Jose Quiles Sebastian - Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SPU.MJQS.SFG.24; FPU22/03291 (Other Grant/Funding Number: Spanish Ministry of Universities)
Record Dates: First submitted 2025-07-09; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Body Esteem

STUDY DESIGN:
Intervention Model Description: Participants are assigned by cluster (classroom) to either an intervention group receiving the IMPACTREEL programme or a waitlist control group. The study uses a parallel group design.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPACTREEL Intervention Group (Experimental): Participants in this arm will receive the IMPACTREEL programme, a school-based intervention combining social media literacy and third-wave strategies (e.g., mindfulness, self-compassion). The programme consists of 7 weekly 55-minute group sessions delivered during school hours by trained facilitators.
  Interventions: Behavioral: IMPACTREEL programme
- Waitlist Control Group (No Intervention): Participants in this arm will receive no intervention during the study period but will be offered the IMPACTREEL programme after the final 12-month follow-up assessment. They will complete the same assessments as the intervention group at baseline, post-intervention, and 6- and 12-month follow-ups.

INTERVENTIONS:
Behavioral: IMPACTREEL programme — The IMPACTREEL programme is a school-based intervention designed to promote positive body image in adolescents. It combines social media literacy education with third-wave strategies, including mindfulness, self-compassion, and psychological flexibility. The intervention consists of 7 weekly group sessions lasting 55 minutes each, delivered by trained psychologists facilitators during school hours. The content targets appearance ideal internalisation, critical thinking about social media, and healthier body image attitudes.
  Arms: IMPACTREEL Intervention Group

SUMMARY:
Background and study aims Many teenagers feel unhappy with their bodies, which can lead to problems like eating disorders, low self-esteem, and depression. Social media plays an important role in shaping how young people see themselves, often promoting unrealistic beauty standards. This study aims to test the effectiveness of a school-based programme called IMPACTREEL, which teaches adolescents how to critically understand social media and improve their relationship with their body using strategies from third-wave psychological therapies. The goal is to help teenagers feel better about their bodies and reduce the risks of developing mental health problems.

Who can participate? The study is open to first year high-school adolescents who attend selected secondary schools in the province of Alicante (Spain). Participation is voluntary, and both the students and their parents/legal guardians must give consent to take part. Young people showing severe symptoms of eating disorders will not be included, as they may need clinical treatment.

What does the study involve?

Participants will be randomly assigned by classroom to one of two groups:

The intervention group will receive the IMPACTREEL programme, which consists of seven weekly sessions, each lasting 55 minutes, delivered at school by trained facilitators.

The control group will not receive the programme during the study but will be offered it later.

Both groups will be asked to complete a series of questionnaires about body image, social media use, emotional well-being, and quality of life before the programme, after it ends, and again 6 months and 12 months later. These questionnaires are confidential and anonymous.

What are the possible benefits and risks of participating? Participants in the intervention group may learn new skills to help them manage how they feel about their body and how they use social media. These strategies may also help reduce stress and improve emotional well-being.

There are no known risks of taking part in this study. Completing the questionnaires or discussing body image may make some students feel uncomfortable, but they are free to stop participating at any time. No clinical diagnosis or treatment is involved in this study.

Where is the study run from? The study is being run by psychologists and researchers from the Universidad Miguel Hernández de Elche (Spain), in collaboration with local secondary schools in the province of Alicante.

When is the study starting and how long is it expected to run for? The study started in 2024 and is expected to continue until 2028, including follow-up assessments and data analysis.

Who is funding the study? The study is funded by a FPU (Formación del Profesorado Universitario) grant from the Spanish Ministry of Universities, which supports doctoral training and research.

Who is the main contact?

Main contact:

Sheila Fernández García Email: sheila.fernandezg@umh.es Affiliation: Universidad Miguel Hernández de Elche

ELIGIBILITY:
Inclusion Criteria:

- Firts year of high-school.

Exclusion Criteria:

- Presence of severe symptoms of eating disorders, indicated by a score above 20 on the EAT-26

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in body esteem | Baseline, post-intervention (week 9), 6-month follow-up, and 12-month follow-up
  Body esteem will be assessed using one validated questionnaire: the Body Esteem Scale for Adolescents and Adults (BESAA). This tool assesses self-perception and satisfaction with one's own body appearance, weight, and attribution by others.
  Body self-esteem measures a person's satisfaction or dissatisfaction with his or her own body. The positive appearance and negative appearance subscales assess overall satisfaction or dissatisfaction with physical appearance, including various visual aspects without focusing on a specific ideal. An example item is: "I like the way I look in pictures". The third subscale, weight, focuses on the person's satisfaction with his or her own weight, as in the item: "I am satisfied with my weight".
  The higher the score, the higher the body esteem. The range of scores is from 18 to 90.

SECONDARY OUTCOMES:
Change in self-compassion | Baseline, post-intervention (week 9), 6-month follow-up, and 12-month follow-up
  Self-compassion will be measured using the Self-Compassion Scale - Youth Version (SCS-Y), which assesses adolescents' ability to treat themselves with kindness and understanding during difficult experiences, particularly those related to body image.
  This instrument measures the degree to which young people respond to their own mistakes and difficulties with kindness, understanding and a balanced perspective. It assesses the ability to treat oneself with understanding in the face of mistakes, measures the ability to recognize imperfections are part of the human experience and the tendency to become angry with oneself when one's own expectations are not met.
  The higher the score, the higher the self-compassion. The range of scores is from 17 to 85.
Change in perceived pressure and comparison on social media | Baseline, post-intervention, 6-month follow-up, 12-month follow-up
  This outcome will be assessed using the Sociocultural Attitudes Towards Appearance Questionnaire -3, Media, Spanish (SATAQ-3-M-S), which evaluates perceived pressure to conform to beauty ideals and the tendency to compare one's appearance with that of celebrities and influencers seen on social media.
  This variable measures the influence of social media on body satisfaction. It measures exposure to content about beauty and body ideals on social media; assesses perceived social pressure to conform to certain appearance standards; and internalization of general beauty ideals related to the body on social media (e.g., being athletic or thin).
  A higher score indicates greater perceived pressure on body image from social media. The score range is from 17 to 85.
Change in internalisation of appearance ideals (SATAQ-4) | Baseline, post-intervention (week 9), 6-month follow-up, and 12-month follow-up
  Internalisation of cultural beauty standards will also be measured using the Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4), which assesses pressure and awareness of appearance norms from media and peers.
  This instrument measures the degree of acceptance of cultural standards of beauty and physical appearance. It assesses the perceived pressure from family, friends, and the media to conform to ideals of thinness, and measures the degree to which the person accepts and pursues the ideal of thinness and the importance of having an athletic and muscular body.
  A higher score indicates greater internalization of the slim and muscular ideal. The score range is from 22 to 110.
Change in social media literacy | Baseline, post-intervention, 6-month follow-up, 12-month follow-up
  Social media literacy will be assessed using a 9 item from three validated measures.
  Items 1-7 were adapted from Tamplin et al. (2018), based on the Critical Thinking about Media Messages Questionnaire (Scull et al., 2010), reworded to reference social media. Item 8 ("I think that physical appearance can only be achieved with filters or editing") was taken from the Fake subscale of the Critical Processing of Beauty Images Scale (Petrie et al., 2019). Item 9 ("People (in real life) look like social media models/influencers") was adapted from the Realism subscale of the Media Attitudes Questionnaire
  Participants rated the frequency of each behaviour on a 6-point Likert scale (1 = never to 6 = always). The higher the score, the greater the social media literacy. The score ranged from 9 to 54.
Change in social media engagement | Baseline, post-intervention, 6-month follow-up, 12-month follow-up
  Social media use will be measured using the Social Media Engagement Scale for Adolescents (SMES-A), which evaluates the frequency, habits, and engagement levels of adolescents with social media platforms.
  This instrument assesses the degree of emotional and behavioural involvement of adolescents with social media, as well as their dependence on it for personal satisfaction and social connection. The items reflect different aspects of social media use, from the habit of constantly checking it to the social reinforcement of using it and the preference for being on social media rather than interacting face to face.
  The higher the score, the greater the engagement with social media. The score ranged from 15 to 75.
Change in eating disorder | Baseline, post-intervention, 6-month follow-up, 12-month follow-up
  Eating disorder risk will be assessed using the Eating Attitudes Test-26 (EAT-26), a screening tool to detect attitudes and behaviours associated with eating disorders.
  The EAT-26 is a questionnaire used to identify eating behaviours and attitudes that may be associated with a risk of developing eating disorders, such as anorexia nervosa (AN) and bulimia nervosa (BN).
  The higher the score, the greater the symptoms of eating disorders. The cut-off point for considering a person at risk is 20 points or more.
Change in depressive symptoms | Baseline, post-intervention, 6-month follow-up, 12-month follow-up
  Depression will be measured using the depression subscale of the Revised Child Anxiety and Depression Scale (RCADS), which assesses symptoms of low mood and emotional distress in young people.
  The subscale measures depressive symptoms in children and adolescents using 10 items that explore various manifestations of sadness, lack of interest, sleep problems, low energy, and feelings of worthlessness. Each item has response options that reflect the frequency of symptoms.
  The higher the score, the greater the depressive symptoms. The score range varies from 0 to 30 points.
Change in life satisfaction | Baseline, post-intervention, 6-month follow-up, 12-month follow-up
  Life satisfaction will be measured using the Satisfaction With Life Scale (SWLS), a five-item measure assessing overall perceived well-being and satisfaction with life.
  A comprehensive measure of personal satisfaction, designed to assess individuals' subjective judgement of their well-being and fulfilment of personal goals. It consists of five items, in which students rate key aspects of their lives, such as achievements, circumstances and overall satisfaction.
  The higher the score, the greater the satisfaction with life. The score range varies from 5 to 25 points.
Change in body image perception | Baseline, post-intervention (week 9), 6-month follow-up, and 12-month follow-up.
  Body image perception will be assessed using the Childress Contour Drawing Rating Scale, a validated figure rating scale that evaluates perceived and ideal body size. Participants select images that represent how they see themselves and how they would like to look, allowing for the assessment of body dissatisfaction.
  To analyse this instrument, the difference in absolute value between the actual body number they consider themselves to have and the ideal body number they would prefer to have is taken into account. If there is no difference, the person is considered to be satisfied with their body. If there is a difference of one or more points between these two items, there will be body dissatisfaction. The greater the difference in score, the greater the body dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: María José Quiles Sebastián María José Quiles Sebastián, Associate Professor, Principal Investigator — Universidad Miguel Hernández de Elche
Locations (1):
- Universidad Miguel Hernández de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected during the trial will be pseudo-anonymised and stored securely in accordance with data protection regulations (GDPR and Spanish data protection law). IPD will not be made publicly available to protect participant confidentiality, particularly due to the involvement of minors. However, de-identified and aggregated data may be made available upon reasonable request to the principal investigator, subject to ethical approval and data-sharing agreements.